CLINICAL TRIAL: NCT01324739
Title: B-type Natriuretic Peptide Affects the Initial Response to Intravenous Glucose in a Placebo-controlled Cross-over Study in Healthy Volunteers
Brief Title: B-type Natriuretic Peptide and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Medical University of Vienna, Department of Endocrinology and Metabolics
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: OeNB 13583
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus; Cardiomyopathy
MeSH Terms: conditions — Diabetes Mellitus; Cardiomyopathies | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B-type natriuretic peptide (Active Comparator): the effect of B-type natriuretic peptide on glucose metabolism will be compared with placebo during an intravenous glocose tolerance test
  Interventions: Drug: human BNP-32
- Placebo (Placebo Comparator): comparison of the effect of b-type natriuretic peptide on glucose metabolism and placebo
  Interventions: Drug: human BNP-32

INTERVENTIONS:
Drug: human BNP-32 — 3pmol/kg/min infusion
  Other Names: human b-type natriuretic peptide

SUMMARY:
Rationale: B type natriuretic peptide (BNP) is a hormone released from cardiomyocytes in response to myocyte stretching and serves as a reliable biomarker in the diagnosis of cardiac dysfunction and heart failure. Recent observations speak for a distinct connection between chronic heart failure and diabetes mellitus.

Objective: The study was set out to investigate the role of BNP on parameters of glucose metabolism in a placebo controlled cross-over study in healthy volunteers.

Methods and Results: Ten participants (25±1 years; BMI 23±1 kg/m2; fasting glucose 83±2 mg/dL) received either placebo or 3 pmol/kg/min BNP 32 intravenously for 4h. One hour after beginning the BNP/placebo infusion, a 3h intravenous glucose tolerance test (0.33 g/kg glucose + 0.03 U/kg insulin at 20 min) was performed and plasma glucose, insulin and C peptide were frequently measured. BNP increased the initial glucose distribution volume (13±1 %BW vs. 11±1, P<0.002), leading to an overall reduction of glucose concentration (P<0.001) especially during the initial 20 min of the test (P=0.001), accompanied by a reduction of the initial C peptide levels (4.3±0.4 ng/mL vs. 4.9±0.3, P=0.015). BNP had no impact on beta cell function, insulin clearance or insulin sensitivity.

Discussion: Intravenous administration of BNP increases glucose initial distribution volume and lowers plasma glucose concentrations after a glucose load without affecting beta cell function or insulin sensitivity what speaks for the concept that BNP is not diabetogenic, but improves the metabolic status in patients with heart failure. This opens new questions regarding BNP induced differences in glucose availability and signalling in several organs/tissues.

DETAILED DESCRIPTION:
In one of our recent studies we investigated insulin sensitivity (OGIS index) and insulin secretion (beta cell function with the insulinogenic index, IGI) in patients with heart insufficiency by frequently sampled oral glucose tolerance test (21). Insulin sensitivity was impaired in CHF compared to control (OGIS: 354±14 ml/min/m2 vs. 450±20; p<0.003). Also beta cell function was reduced (IGI: 100±14 vs. 150±45 pmolINS/pmolGLUC). Interestingly a significant inverse correlation exists between BNP and IGI (r=0.41, p<0.05) (21). The relationship between BNP and glucose metabolism has only been partially investigated. Plasma BNP rises in response to hyperglycemia, but is not influenced by hyperinsulinemia (22, 23). On the other side, the physiological role of BNP on beta cell function and insulin sensitivity has not been investigated to date. As BNP levels rise with the degree of heart insufficiency and insulin resistance correlates to the degree of cardiomyopathy, we hypothesize that BNP influences glucose metabolism in healthy men.

One gold standard investigation of both beta cell function and peripheral insulin sensitivity is the insulin-modified frequently sampled intravenous glucose tolerance test (FSIGT). The FSIGT consists in giving intravenously a glucose bolus at time point 0 followed by an intravenous administration of insulin at time point 20 minutes (18,19, 20). The determination of glucose, insulin and C-peptide at frequent intervals till time point 180 minutes allows the calculation of the acute insulin response, glucose effectiveness, insulin clearance and insulin sensitivity through the minimal model analysis (13) The intravenous administration of 3 pmol/kg/min BNP achieves a plateau of increased BNP plasma concentrations after 60 minutes. In previous publications, this infusion was administered during 4 hours, achieving a steady state plasma BNP between time points 60 minutes and 240 minutes (17). Using this already established protocol, we aim to maintain constantly high plasma BNP levels throughout the three hours of the FSIGT. The combination of both BNP (17) and FSIGT (13) protocols in an interventional study will be an adequate means of investigating the impact of BNP on glucose metabolism in healthy subjects.

The present study aims to investigate the effect of intravenous infusion of BNP-32 (American Peptide, Calif., US) on the beta cell function and insulin sensitivity during FSIGT in healthy volunteers.

-65, -60, -30, 0, 3, 4, 5, 6, 8, 10, 14, 19, 22, 27, 30, 35, 40, 50, 60, 70, 90, 100, 120, 140, 150 and 180 min for the measurement of glucose, insulin and C-peptide (8 ml per time point: time points -30, 0, 3, 4, 5, 6, 8, 10, 14, 19, 22, 27, 30, 35, 40, 50, 70, 100, 140 and 180 min), for the measurement of BNP and NT-proBNP (4 ml per time point: time points -65, -60, -30, 0, 30, 60, 90, 120, 150 and 180 min) and for the measurement of plasma sodium, potassium and creatinine (8 ml per time point: time points -60, 60 and 180 minutes).

Primary outcome parameter is area under the curve of insulin (AUCinsulin) from time point -30 to 180 min.

Secondary outcome parameters are AUCglucose and AUCc-peptide from time point -30 to 180 min, BNP- and NT-proBNP levels from time point -65 to 180, plasma sodium, potassium and creatinine from time point -60 to 180.

On study days volunteers will come to the study room at around 07:45 a.m. after an overnight fasting. After being weighed, they will remain in bed throughout the study, except when standing to pass urine. Two vein flow needles (Venflon, Helsingborg, Sweden) will be inserted in the antecubital veins of the right and left arm for the administration of infusions and blood sampling respectively. The subjects will rest for approximately 15 minutes before obtaining baseline blood samples (at time point - 65 minutes).

3.0 pmol/kg/min human BNP-32 (American Peptide, Calif., US) which is solved in Haemaccel (10 mL/h), or placebo (Haemaccel, 10 mL/h, alone) will be continuously administered for 4 hours, between time points -60 and 180 minutes, using a syringe pump (Treonic, Vickers Medical, Basingstoke, United Kingdom). A washout period of at least 2 weeks will be between the administration of BNP and placebo on the two different study days. This protocol has been used in the study of Lainchbury et al. (17).

330 mg/kg body weight glucose will be administered as a bolus during 30 seconds at time point 0-0.5 minutes.

0.03 IU/kg rapidly acting insulin (Actrapid, Novo-Nordisk, Denmark) will be infused intravenously for 5 minutes starting at time point 20.

Blood samples will be collected at time points: -65, -60, -30, 0, 3, 4, 5, 6, 8, 10, 14, 19, 22, 27, 30, 35, 40, 50, 60, 70, 90, 100, 120, 140, 150 and 180 min for the measurement of glucose, insulin and C-peptide (8 ml per time point: time points -30, 0, 3, 4, 5, 6, 8, 10, 14, 19, 22, 27, 30, 35, 40, 50, 70, 100, 140 and 180 min), for the measurement of BNP and NT-proBNP (4 ml per time point: time points -65, -60, -30, 0, 30, 60, 90, 120, 150 and 180 min) and for the measurement of plasma sodium, potassium and creatinine (8 ml per time point: time points -60, 60 and 180 minutes).

A final safety blood sample will be collected at time point 270 min for plasma sodium, potassium, creatinine and BNP, NT-proBNP, sodium, potassium, creatinine, GPT, gamma-GT, total bilirubin to ensure that (NT-pro)BNP levels returned to baseline and other parameters are within the normal range.

Total volume of blood withdrawal will be about 230 ml. When voiding, the subjects will be asked to collect the urine excreted during the study period (-65 till 180 minutes). for the measurement of sodium, potassium and creatinine excretion.

Heart rate and blood pressure will be continuously monitored during the whole study. If the systolic blood pressure is lower than 85 mmHg or the heart rate is less than 50 beats per minute BNP infusion will be stopped.

Data analysis for estimating insulin sensitivity, ß-cell secretion, insulin clearance, insulin hepatic extraction and insulin appearance rate will be done by minimal model computer analysis of the frequently sampled intravenous glucose tolerance test

ELIGIBILITY:
Inclusion Criteria:

written informed consent no disease history BNP level within the normal range Normal renal function (serum creatinine of more than 1.3 mg/dL and/or creatinin clearance greater than 80ml/min) Normal ECG

Exclusion Criteria:

systolic blood pressure < 90 mmHg subjects on any medication abnormal glucose metabolism history of anaphylaxis

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
glucose | 0 to 180 minutes

SECONDARY OUTCOMES:
insulin, c-peptide | 0 to 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clodi, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Heinisch BB, Vila G, Resl M, Riedl M, Dieplinger B, Mueller T, Luger A, Pacini G, Clodi M. B-type natriuretic peptide (BNP) affects the initial response to intravenous glucose: a randomised placebo-controlled cross-over study in healthy men. Diabetologia. 2012 May;55(5):1400-5. doi: 10.1007/s00125-011-2392-1. Epub 2011 Dec 13. PMID 22159910